CLINICAL TRIAL: NCT03533933
Title: Clinical and Histomorphometric Analysis of Collagen Matrix Versus Connective Tissue Graft in Mucogingival Surgery in Orthodontic Patients. A Randomized, Controlled Clinical Trial
Brief Title: Clinical and Histomorphometric Analysis of Collagen Matrix Versus Connective Tissue Graft in Mucogingival Surgery in Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elena Ruiz de Gopegui Palacios (Other)
Responsible Party: Sponsor-Investigator, Elena Ruiz de Gopegui Palacios, Principal investigator, University of the Basque Country (UPV/EHU)
Organization: University of the Basque Country (UPV/EHU) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCP-2
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Gingival Recession
Keywords: collagen matrix; connective tissue graft; histometry; xenograft; periodontal regeneration; biometry
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Split mouth
Who Masked: Outcomes Assessor
Masking Description: Analyst and Histometry: The statistician and the pathologist does not know which treatment corresponds to each variable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous connective tissue graft (Active Comparator): Soft tissue harvesting from patient palate
  Interventions: Other: autologous connective tissue graft
- collagen matrix (Experimental): Mucograft collagen matrix manufactured by Geistlich AG, Switzerland Device: Collagen matrix
  Interventions: Device: Collagen matrix

INTERVENTIONS:
Device: Collagen matrix — Mucograft collagen matrix combined with coronal advanced flap
  Arms: collagen matrix
Other: autologous connective tissue graft — Soft tissue harvesting from patient palate with coronal advanced flap
  Arms: Autologous connective tissue graft

SUMMARY:
There are some orthodontics treatments that perform risk movements ,and a bone dehiscence may be expected. In that cases mucogingival surgery , such as connective tissue grafts, is necessary prior to tooth movement.

The connective tissue graft in combination with coronal advanced flap is still considered the gold standard , although the use of porcine collagen matrix has obtained promising results for treatment of Miller class I and II recession defects.

Most of the studies report clinical results after a connective tissue graft and there is no evidence about the type of attachment obtained after the graft is performed, a few articles have shown histological results. But, as a rule , a histological study is only performed under exceptional circumstances such as a dental fracture, untreatable decay, tooth extraction for orthodontic reasons, or other reasons.

Most of the techniques results in the formation of a long junctional epithelium and connective tissue attachment with fibers parallel to the root surface. Animals studies have shown a shorter epithelium and a larger new cementum formation after the use of the collagen matrix.

DETAILED DESCRIPTION:
The purpose of this study is to confirm that periodontal regeneration happens after mucogingival surgery The principal outcome is compare the millimeters of new attachment create after a connective tissue graft and after the use of a porcine collagen matrix in teeth that have to been extracted (because of the orthodontic planing treatment) after mucogingival surgery .

The secondary outcomes are:

1. length of new cementum (histometry results)
2. length of the junctional epithelium (histometry results)
3. length of connective tissue attachment (histometry results)
4. complete root coverage (clinical results)
5. width of keratinized tissue

ELIGIBILITY:
Inclusion Criteria:

* Patient in orthodontic treatment ,who needs mucogingival surgery in both hemi arcade and later the tooth adjacent to the graft should be extracted because of the orthodontic planing treatment .
* The patient must be 18 years or older
* Patient shows sufficient plaque control (FMPS < 20%).
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent

Exclusion Criteria:

* General contraindications for dental and/or surgical treatment are present.
* The patient is taking medications or having treatments which have an effect on mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs).
* Untreated periodontal conditions
* Patients not willing to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
millimeters of new attachment | Change from baseline at following surgery sixth month
  histometry assessment

SECONDARY OUTCOMES:
Length of new cementum | Change from baseline at following surgery sixth month
  histometry assessment
Length of new junctional epithelium | Change from baseline at following surgery sixth month
  histometry assessment
length of connective attachment | Change from baseline at following surgery sixth month
  histometry assessment
complete root coverage | Change from baseline at following surgery sixth month
  clinical assessment
width of keratinized tissue | Change from baseline at following surgery sixth month
  clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Luis Antonio Aguirre Zorzano, Study Director — University of the Basque Country (UPV/EHU); Elena Ruiz de Gopegui, Principal Investigator — University of the Basque Country (UPV/EHU); Ana Maria Garcia de la Fuente, Principal Investigator — University of the Basque Country (UPV/EHU); Ruth Estefania Fresco, Study Chair — University of the Basque Country (UPV/EHU); Xavier Marichalar Mendia, Study Chair — University of the Basque Country (UPV/EHU); Jose Manuel Aguirre Urizar, Study Chair — University of the Basque Country (UPV/EHU)
Locations (1):
- Department fo Stomatology II, Faculty of Medicine and Nursery, University of the Basque Country, Leioa, Biscay, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data collected for the study will be identified by a code and only the researcher will be able to relate them. The personal data will be treated with absolute confidentiality in accordance with the Data Protection Law and will remain in the patient's clinical history. The coded data will be included in a UPV/EHU´s file with reference number 2080310015-INA0110, whose head is Ana María García de la Fuente, and will only be used for the purposes of this project.

REFERENCES:
- [Background] Batenhorst KF, Bowers GM, Williams JE Jr. Tissue changes resulting from facial tipping and extrusion of incisors in monkeys. J Periodontol. 1974 Sep;45(9):660-8. doi: 10.1902/jop.1974.45.9.660. No abstract available. PMID 4529575
- [Background] Steiner GG, Pearson JK, Ainamo J. Changes of the marginal periodontium as a result of labial tooth movement in monkeys. J Periodontol. 1981 Jun;52(6):314-20. doi: 10.1902/jop.1981.52.6.314. PMID 6943326
- [Background] Wennstrom JL, Lindhe J, Sinclair F, Thilander B. Some periodontal tissue reactions to orthodontic tooth movement in monkeys. J Clin Periodontol. 1987 Mar;14(3):121-9. doi: 10.1111/j.1600-051x.1987.tb00954.x. PMID 3470318
- [Background] Buti J, Baccini M, Nieri M, La Marca M, Pini-Prato GP. Bayesian network meta-analysis of root coverage procedures: ranking efficacy and identification of best treatment. J Clin Periodontol. 2013 Apr;40(4):372-86. doi: 10.1111/jcpe.12028. Epub 2013 Jan 24. PMID 23346965
- [Background] Cairo F, Pagliaro U, Nieri M. Treatment of gingival recession with coronally advanced flap procedures: a systematic review. J Clin Periodontol. 2008 Sep;35(8 Suppl):136-62. doi: 10.1111/j.1600-051X.2008.01267.x. PMID 18724847
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Background] Thoma DS, Benic GI, Zwahlen M, Hammerle CH, Jung RE. A systematic review assessing soft tissue augmentation techniques. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:146-65. doi: 10.1111/j.1600-0501.2009.01784.x. PMID 19663961
- [Background] Thoma DS, Muhlemann S, Jung RE. Critical soft-tissue dimensions with dental implants and treatment concepts. Periodontol 2000. 2014 Oct;66(1):106-18. doi: 10.1111/prd.12045. PMID 25123764
- [Background] Soileau KM, Brannon RB. A histologic evaluation of various stages of palatal healing following subepithelial connective tissue grafting procedures: a comparison of eight cases. J Periodontol. 2006 Jul;77(7):1267-73. doi: 10.1902/jop.2006.050129. PMID 16805692
- [Background] Griffin TJ, Cheung WS, Zavras AI, Damoulis PD. Postoperative complications following gingival augmentation procedures. J Periodontol. 2006 Dec;77(12):2070-9. doi: 10.1902/jop.2006.050296. PMID 17209793
- [Background] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Treatment of gingival recession defects using coronally advanced flap with a porcine collagen matrix compared to coronally advanced flap with connective tissue graft: a randomized controlled clinical trial. J Periodontol. 2012 Mar;83(3):321-8. doi: 10.1902/jop.2011.110215. Epub 2011 Jul 1. PMID 21721988
- [Background] Aroca S, Molnar B, Windisch P, Gera I, Salvi GE, Nikolidakis D, Sculean A. Treatment of multiple adjacent Miller class I and II gingival recessions with a Modified Coronally Advanced Tunnel (MCAT) technique and a collagen matrix or palatal connective tissue graft: a randomized, controlled clinical trial. J Clin Periodontol. 2013 Jul;40(7):713-20. doi: 10.1111/jcpe.12112. Epub 2013 Apr 30. PMID 23627374
- [Background] Jepsen K, Jepsen S, Zucchelli G, Stefanini M, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M. Treatment of gingival recession defects with a coronally advanced flap and a xenogeneic collagen matrix: a multicenter randomized clinical trial. J Clin Periodontol. 2013 Jan;40(1):82-9. doi: 10.1111/jcpe.12019. Epub 2012 Oct 10. PMID 23050490
- [Background] Molnar B, Aroca S, Keglevich T, Gera I, Windisch P, Stavropoulos A, Sculean A. Treatment of multiple adjacent Miller Class I and II gingival recessions with collagen matrix and the modified coronally advanced tunnel technique. Quintessence Int. 2013 Jan;44(1):17-24. doi: 10.3290/j.qi.a28739. PMID 23444157
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Coronally advanced flap with and without a xenogenic collagen matrix in the treatment of multiple recessions: a randomized controlled clinical study. Int J Periodontics Restorative Dent. 2014;34 Suppl 3:s97-102. doi: 10.11607/prd.1605. PMID 24956099
- [Background] Atieh MA, Alsabeeha N, Tawse-Smith A, Payne AG. Xenogeneic collagen matrix for periodontal plastic surgery procedures: a systematic review and meta-analysis. J Periodontal Res. 2016 Aug;51(4):438-52. doi: 10.1111/jre.12333. Epub 2015 Nov 7. PMID 26547393
- [Background] McGuire MK, Scheyer ET. Long-Term Results Comparing Xenogeneic Collagen Matrix and Autogenous Connective Tissue Grafts With Coronally Advanced Flaps for Treatment of Dehiscence-Type Recession Defects. J Periodontol. 2016 Mar;87(3):221-7. doi: 10.1902/jop.2015.150386. Epub 2015 Oct 15. PMID 26469812
- [Result] Harris RJ. Successful root coverage: a human histologic evaluation of a case. Int J Periodontics Restorative Dent. 1999 Oct;19(5):439-47. PMID 10709509
- [Result] Carnio J, Camargo PM, Kenney EB. Root resorption associated with a subepithelial connective tissue graft for root coverage: clinical and histologic report of a case. Int J Periodontics Restorative Dent. 2003 Aug;23(4):391-8. PMID 12956483
- [Result] Pasquinelli KL. The histology of new attachment utilizing a thick autogenous soft tissue graft in an area of deep recession: a case report. Int J Periodontics Restorative Dent. 1995 Jun;15(3):248-57. PMID 7558658
- [Result] Bruno JF, Bowers GM. Histology of a human biopsy section following the placement of a subepithelial connective tissue graft. Int J Periodontics Restorative Dent. 2000 Jun;20(3):225-31. PMID 11203564
- [Result] Goldstein M, Boyan BD, Cochran DL, Schwartz Z. Human histology of new attachment after root coverage using subepithelial connective tissue graft. J Clin Periodontol. 2001 Jul;28(7):657-62. doi: 10.1034/j.1600-051x.2001.028007657.x. PMID 11422587
- [Result] Majzoub Z, Landi L, Grusovin MG, Cordioli G. Histology of connective tissue graft. A case report. J Periodontol. 2001 Nov;72(11):1607-15. doi: 10.1902/jop.2001.72.11.1607. PMID 11759874
- [Result] Garcia-De-la-Fuente AM, Aguirre-Zorzano LA, Estefania-Fresco R, Roig Odena L, Aguirre-Urizar JM. Histologic and Clinical Study of Gingival Recession Treated with Subepithelial Connective Tissue Graft: A Case Report. Int J Periodontics Restorative Dent. 2017 Jan/Feb;37(1):89-97. doi: 10.11607/prd.2638. PMID 27977823
- [Result] McGuire MK, Nunn M. Evaluation of human recession defects treated with coronally advanced flaps and either enamel matrix derivative or connective tissue. Part 1: Comparison of clinical parameters. J Periodontol. 2003 Aug;74(8):1110-25. doi: 10.1902/jop.2003.74.8.1110. PMID 14514224
- [Result] Roman A, Campian R, Domsa I, Soanca A, Gocan H. Subepithelial connective tissue graft for root coverage: clinical case reports and histologic evaluation. Rom J Morphol Embryol. 2010;51(4):793-7. PMID 21103645
- [Result] Harris RJ. Root coverage with a connective tissue with partial thickness double pedicle graft and an acellular dermal matrix graft: a clinical and histological evaluation of a case report. J Periodontol. 1998 Nov;69(11):1305-11. doi: 10.1902/jop.1998.69.11.1305. PMID 9848542